CLINICAL TRIAL: NCT06984328
Title: Efficacy and Safety Study of Acasunlimab as Monotherapy and in Combination With Pembrolizumab in Subjects With Relapsed/Refractory, Unresectable Locally Advanced or Metastatic Cutaneous Melanoma That Progressed On or After Treatment With a Checkpoint Inhibitor (ABBIL1TY MELANOMA-07)
Brief Title: Study of the Effectiveness and Safety of Acasunlimab Alone and With Pembrolizumab to Treat Advanced Melanoma of the Skin That Has Returned After Treatment With an Approved Checkpoint Inhibitor Therapy (ABBIL1TY MELANOMA-07)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1046-07; 2025-520468-16 (Other: EU CT No.)
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous Melanoma; Relapsed/Refractory, Locally Advanced Unresectable Melanoma (Stage IIIB, IIIC, or IIID); Metastatic Cutaneous Melanoma (Stage IV)
Keywords: Melanoma; Cutaneous Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Acasunlimab in Combination with Pembrolizumab (Experimental): Participants with relapsed/refractory, unresectable locally advanced or metastatic cutaneous melanoma that progressed on/after prior CPI(s) will receive acasunlimab once every 6 weeks (Q6W) in combination with pembrolizumab Q6W.
  Interventions: Biological: Acasunlimab; Biological: Pembrolizumab
- Acasunlimab (Experimental): Participants with relapsed/refractory, unresectable locally advanced or metastatic cutaneous melanoma that progressed on/after prior CPI(s) will receive acasunlimab Q6W.
  Interventions: Biological: Acasunlimab

INTERVENTIONS:
Biological: Acasunlimab — Intravenous (IV) infusion
  Other Names: GEN1046; DuoBody®-PD-L1×4-1BB
Biological: Pembrolizumab — IV infusion
  Arms: Acasunlimab in Combination with Pembrolizumab

SUMMARY:
The goal of this clinical trial is to learn about the effectiveness and safety of the bispecific antibody acasunlimab (also known as DuoBody®-PD-L1x4-1BB) when given either alone or together with the cancer drug pembrolizumab in participants with locally advanced or metastatic melanoma of the skin. All participants will receive active drugs; no one will be given a placebo.

The trial duration will be approximately 15 months for each participant, including a 28-day screening period and estimated 4-month treatment and 10-month follow-up periods; however, the duration of the treatment and follow-up periods may vary for each participant.

Participants will have regular check-ups while on treatment, with visits every week initially, and then every 3 weeks later in the trial.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, open-label, multicenter trial evaluating the efficacy and safety of acasunlimab as monotherapy and in combination with pembrolizumab in adult participants with relapsed/refractory, unresectable locally advanced or metastatic cutaneous melanoma who progressed on or after prior checkpoint inhibitor (CPI)-containing therapy. Participants will be randomized in a 1:1 ratio to receive acasunlimab and pembrolizumab or acasunlimab alone.

Eligible participants must have received a minimum of 2 cycles of an approved anti-programmed cell death protein 1 (PD-1) containing therapy. Participants whose tumor harbors a B-Raf proto-oncogene, serine/threonine kinase (BRAF) V600 mutation are eligible for the trial if they have received a BRAF-directed therapy (with or without a mitogen-activated protein kinase [MEK] inhibitor) prior to enrollment in the trial, unless the investigator has deemed a BRAF-directed therapy not clinically indicated. BRAF V600 mutational status must be determined by local assessment and documented.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants ≥ 18 years of age with histologically or cytologically confirmed diagnosis of relapsed/refractory, locally advanced unresectable (Stage IIIB, IIIC, or IIID) or metastatic (Stage IV) cutaneous melanoma, per American Joint Committee on Cancer (8th edition) staging.
* Participant must have radiographic progression based on RECIST v1.1 on or following ≥ 1 prior systemic therapy, according to local and international guidelines, including a programmed cell death protein 1 blocking antibody (anti-PD-1) treatment or combination treatment containing an anti-PD-1.
* Participant must have received a minimum of 2 cycles of an approved anti-PD-1 as monotherapy or a combination therapy containing an anti-PD-1.
* Neoadjuvant and/or adjuvant systemic therapy count as the first line of prior systemic therapy if there is documented disease progression ≤ 6 months after completion of therapy.
* Participants with a BRAF V600 mutation should have received prior BRAF-directed therapy (with or without a MEK inhibitor) prior to enrollment in the trial, unless deemed not clinically indicated by the Investigator due to concurrent medical condition or prior toxicity.
* Participant has an Eastern Cooperative Oncology Group performance status of 0 or 1 within 7 days prior to Cycle 1 Day 1.

Key Exclusion Criteria:

* Participants with non-cutaneous or acral melanoma.
* Participants with newly identified or known unstable or symptomatic central nervous system metastases or history of carcinomatous meningitis.

Note: Other protocol-defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-07-25 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  Assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Time to Response (TTR) | Up to approximately 15 months
  Assessed by the investigator per RECIST v1.1.
Duration of Response (DOR) | Up to approximately 15 months
  Assessed by the investigator per RECIST v1.1.
Progression-free Survival (PFS) | Up to approximately 15 months
  Assessed by the investigator per RECIST v1.1.
Overall Survival (OS) | Up to approximately 15 months
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 15 months
Time to Treatment Discontinuation Due to Adverse Events (AEs) | Up to approximately 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (2):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States
- Pan American Center for Oncology Trials, LLC, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No